CLINICAL TRIAL: NCT03167736
Title: The Addition of Electric Dry Needling and Spinal Manipulation to Impairment-based Manual Therapy, Stretching, Strengthening and Electrothermal Modalities for Patients With Lumbar Spinal Stenosis: a Multi-randomized Clinical Trial
Brief Title: Dry Needling and Spinal Manipulation vs. Conventional PT for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Primary Investigator and President of Spinal Manipulation Institute and Dry Needling Institute of the American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0011
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric dry needling, manipulation (Experimental)
  Interventions: Other: electric dry needling, manipulation
- conventional physical therapy (Active Comparator)
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: electric dry needling, manipulation — HVLA thrust manipulation to lumbar spine. Dry needling to lumbar/sacral paraspinal muscles and gluteus medium/minimus muscles. Treatment may include dry needling of the piriformis muscle, quadrates lumborum muscle and perineurial needling of sciatic/tibial nerve. Up to 12 treatment sessions over 6 weeks.
  Arms: Electric dry needling, manipulation
Other: conventional physical therapy — Impairment-based manual therapy, stretching, strengthening and electrothermal modalities targeting the lumbar/sacral spine and hips. Up to 12 treatment sessions over 6 weeks.
  Arms: conventional physical therapy

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with lumbar spinal stenosis: electric dry needling and thrust manipulation versus impairment-based manual therapy, stretching, strengthening and electrothermal modalities. Physical therapists commonly use all of these techniques to treat lumbar spinal stenosis. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with lumbar spinal stenosis will be randomized to receive 1-2 treatment sessions per week for 6 weeks (up to 12 sessions total) of either: (1) electric dry needling and thrust manipulation or (2) impairment-based manual therapy, stretching, strengthening and electrothermal modalities

ELIGIBILITY:
Inclusion Criteria:

1. Adult over the age of 50 years old that is able to read, write and speak English
2. Symptoms of neurogenic claudication (pain in the buttock, thigh, or leg during ambulation that improves with rest) or radicular leg symptoms with associated neurological deficits on the physical examination for at least 12 weeks.
3. Confirmatory imaging (i.e. magnetic resonance imaging (MRI), computed tomography (CT), myelography, ultrasound or X-ray of either central or lateral (foraminal) lumbar spinal stenosis at one or more levels in the lumbar spine.

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: severe hypertension, infection, ankylosing spondylitis, neoplasm, uncontrolled diabetes, peripheral neuropathy, heart disease, stroke, chronic, ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. Severe vascular, pulmonary, or coronary artery disease limiting participation in exercise, to include a walking program (including presence of absolute contraindications to submaximal exercise testing)
3. Severe degenerative stenosis with intractable pain and progressive neurological dysfunction
4. Lumbar spinal stenosis not caused by degeneration
5. Radiographic evidence of instability, degenerative spondylolisthesis, fracture or scoliosis of more than 15°
6. Lumbar herniated disc diagnosis during the last 12 months.
7. Previous lumbar surgery for lumbar spinal stenosis or instability (i.e. previous lumbar fusion, lumbar microdiscectomy, lumbar foraminotomy, lumbar laminectomy, etc.)
8. Psychiatric disorder or cognitively impaired.
9. Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in low back pain (NPRS) (Rating Score) | baseline, 2-weeks, 6-weeks and 3-months
  Baseline score must exceed 2/10 to be included in the study.
Change in Oswestry Disability Index | baseline, 2-weeks, 6-weeks and 3-months
  The Oswestry Disability Index (ODI) includes 10 questions, each worth 0-5 points with maximum score of 50 points possible. The greater the score, the worse the disability. Baseline score must exceed 10/50 points to be included in the study.

SECONDARY OUTCOMES:
Change in Roland Morris Disability Index | baseline, 2-weeks, 6-weeks and 3-months
  The Roland Morris Disability Index (RMDI) is measured on a 0-24 scale. Greater scores indicate increased disability.
Change in Global Rating of Change Score | 2-weeks, 6-weeks and 3-months
Change in Medication Intake (Frequency of medication intake in last week) | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Benchmark PT - Canton, Canton, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided